CLINICAL TRIAL: NCT00068770
Title: A Pharmacokinetic Study of the Interaction Between Celecoxib and Anticonvulsant Drugs in Patients With Newly Diagnosed Glioblastoma Multiforme Undergoing Radiation Therapy
Brief Title: Celecoxib in Patients With Newly Diagnosed GBM Who Are Receiving Anticonvulsant Drugs and Undergoing RT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: EORTC trail showed TMZ & RT conferred significant survivial in this population
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NABTT-2100 CDR0000328117; U01CA062475 (NIH); NABTT-2100; JHOC-NABTT-2100
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Radiotherapy; Celecoxib; Cyclooxygenase 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- p450 ( +EIASD) (Active Comparator): on p450 inhibitor (Patients taking anttiseizure drugs that are known to induce the hepatic drug-metabolizing enzymes - including phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine)
  celecoxib and radiation therapy will be adminstered with this arm
  Interventions: Radiation: radiation therapy; Drug: Celecoxib
- nonp450 (-EIASD) (Active Comparator): not on p450 inhibitor (Patients either NOT taking anti-seizure drugs or ones that are known to not significantly influence the hepatic drug-metabolizing enzymes - including gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine,topiramate, zonisamide and filbamate.
  celecoxib and radiation therapy will be adminstered with this arm
  Interventions: Radiation: radiation therapy; Drug: Celecoxib

INTERVENTIONS:
Radiation: radiation therapy — Radiation is standard treatment 6000cGy in 30 fractions. Patients will receive celecoxib 400 mg bid during RT treatment
  Other Names: RT
Drug: Celecoxib — Celecoxib will begin 1 week prior to RT at 400mg bid orally. One day 1 only 1 dose will be administered. Starting on day 2 and throughout treatment until progression, 2 doses will be administered at least 12 hours apart. Celecoxib will continue throughout the 6 week course of RT.
  Other Names: Cox2

SUMMARY:
RATIONALE: Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. It is not yet known whether the effectiveness of celecoxib in treating glioblastoma multiforme is decreased in patients who are receiving anticonvulsant drugs and undergoing radiation therapy.

PURPOSE: Phase II trial to study the effectiveness of celecoxib in treating patients who are receiving anticonvulsant drugs and undergoing radiation therapy for newly diagnosed glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effects of hepatic enzyme-inducing drugs, such as anticonvulsants, on the pharmacokinetics of celecoxib in patients with newly diagnosed glioblastoma multiforme undergoing radiotherapy.
* Determine the effects of steroids on the pharmacokinetics of celecoxib in these patients.

Secondary

* Determine the safety of celecoxib in these patients.
* Determine the duration of survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients are assigned to 1 of 2 groups based on anticonvulsant therapy.

* Group A: Patients treated with any of the following anticonvulsant drugs that induce hepatic metabolic enzymes:

  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Primidone
  * Oxcarbazepine
* Group B: Patients treated with any of the following anticonvulsant drugs that cause modest or no induction of hepatic metabolic enzymes OR no anticonvulsant drug:

  * Gabapentin
  * Lamotrigine
  * Valproic acid
  * Levetiracetam
  * Tiagabine
  * Topiramate
  * Zonisamide
  * Felbamate
* Induction therapy: Patients in both groups receive oral celecoxib twice* daily on weeks 1-11 and undergo radiotherapy 5 days a week on weeks 2-7.
* Maintenance therapy: Patients receive oral celecoxib twice daily. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients receive only 1 dose on the first day of celecoxib administration.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 44 patients (22 per group) will be accrued for this study within approximately 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Supratentorial
  * Grade IV astrocytoma

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* Transaminases no greater than 4 times upper limit of normal

Renal

* Creatinine no greater than 1.7 mg/dL
* Creatinine clearance at least 60 mL/min
* No prior renal toxicity with nonsteroidal anti-inflammatory drugs

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Mini mental score at least 15
* No history of peptic disease
* No serious concurrent infection
* No other medical illness that would preclude study participation
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer
* No allergy to sulfonamides
* Able to tolerate cyclo-oxygenase-2 (COX-2) inhibitors

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy or biologic agents for the malignancy, including any of the following:

  * Immunotoxins
  * Immunoconjugates
  * Antisense agents
  * Peptide receptor antagonists
  * Interferons
  * Interleukins
  * Tumor-infiltrating lymphocytes
  * Lymphokine-activated killer cells
  * Gene therapy
* No concurrent prophylactic growth factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy

* No prior chemotherapy for the malignancy

Endocrine therapy

* No prior hormonal therapy for the malignancy
* Prior glucocorticoid therapy allowed
* Concurrent corticosteroids allowed provided there has been no dose increase within the past 5 days

Radiotherapy

* No prior radiotherapy for the malignancy

Surgery

* Recovered from prior surgery

Other

* At least 1 week since prior fluconazole
* More than 10 days since prior anticonvulsant drugs that induce hepatic metabolic enzymes (Group A)
* No other prior therapy for the malignancy
* No concurrent enrollment in another therapeutic clinical trial
* No concurrent fluconazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-10; Primary Completion 2005-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart A. Grossman, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (7):
- United States (7):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Grossman SA, Olson J, Batchelor T, Peereboom D, Lesser G, Desideri S, Ye X, Hammour T, Supko JG; New Approaches to Brain Tumor Therapy CNS Consortium. Effect of phenytoin on celecoxib pharmacokinetics in patients with glioblastoma. Neuro Oncol. 2008 Apr;10(2):190-8. doi: 10.1215/15228517-2007-055. Epub 2008 Feb 20. PMID 18287342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: pts were enrolled on this study from October 2003 to September 2004. Pts were enrolled in an outpatient clinical setting
Pre-assignment Details: pts were assigned to an arm at the time of enrollment
Groups:
- nonp450: not on p450 inhibitor
  celecoxib :
  radiation therapy :
- p450: on p450 inhibitor
  celecoxib :
  radiation therapy :
Period: Overall Study
Arm/Group | nonp450 | p450
Started | 13 | 22
Completed | 13 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- p450 ( +EIASD): on p450 inhibitor (Patients taking anttiseizure drugs that are known to induce the hepatic drug-metabolizing enzymes - including phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine)
- nonp450 (-EIASD): not on p450 inhibitor (Patients either NOT taking anti-seizure drugs or ones that are known to not significantly influence the hepatic drug-metabolizing enzymes - including gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine,topiramate, zonisamide and filbamate.
- Total: Total of all reporting groups
Arm/Group | p450 ( +EIASD) | nonp450 (-EIASD) | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12) | 56 (17) | 57 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 14 | 6 | 20
Karnofsky Perfomance Status (KPS) [Mean (Standard Deviation); unit: scores on a scale] — 100 normal no complaints no disease 90 capable of normal activity few symptoms/disease 80 normal activity with some difficulty some symptoms or signs 70 caring for self not capable of normal activity or work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care and help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures or treatment 10 moribund rapidly progressive fatal disease processes 0 death
  scores on a scale | 88 (11) | 83 (9) | 86 (10)
Mini Mental State Exam Score [Mean (Standard Deviation); unit: scores on a scale] — The mini-mental state examination (MMSE) is a 30-point questionnaire test used to screen for cognitive impairment. Commonly used to screen for dementia. It is also used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time. The MMSE test includes simple questions and problems in a number of areas: the time and place of the test, repeating lists of words, arithmetic such as the serial sevens, language use and comprehension, and basic motor skills. The Higher your score, the higher your function.
  scores on a scale | 28 (4) | 28 (3) | 28 (3)
Corticosteroid therapy [Number; unit: Participants] — Patients on corticpsteroid therapy
  Participants
    Yes | 18 | 11 | 29
    No | 4 | 2 | 6
Prior Surgery [Number; unit: Participant] — Whether pt had Craniotomy or Biopsy
  Participant
    Craniotomy | 21 | 10 | 31
    Biopsy | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Effects of Hepatic Enzyme Inducing Drugs Such as Anticonvulsants, on the PK of Celecoxib
Description: subjects will take one dose of celecoxib and will then have 6 hours of blood draws, day 2 subject will take 2 doses of celecoxib 8 hours apart with 2 additional blood samples, one hour apart. Subject, will continue to take 2 doses of celecoxib for 6 weeks, with a sample (PK) drawn every week prior to the first dose of the week. Comparison of Cmax of Celecoxib is reported
Time Frame: First dose of celecoxib through completion of radiation, 6 weeks.
Population: pts who had PK data for the first dose of celecoxib. observations were excluded if sample was not collected within 12 +/- 2h after taking prior dose, was drawn after dosing on same day or determine to be outlier by dixon's test.
  PK data was available for 15 pts in the +EIASD group and 12 pts in the -EIASD group
Measure: Geometric Mean (Standard Deviation); unit: (ng/ml)
Arm/Group | nonp450 | p450
Number analyzed (Participants) | 12 | 15
(ng/ml) | 1752 (550) | 1813 (813)
Statistical Analysis 1: Comparison: nonp450 vs p450; two independent group comparisons; Test type: Superiority or Other; p = 0.82, t-test, 2 sided — not adjusted; Mean Difference (Final Values) = 3.5, 95% CI 2-sided [1.5 to 5.5], Standard Deviation 1

2. Secondary Outcome: Overall Survival
Description: duration of survival when celecoxib is administered concurrently with radiation in pts with newly diagnosed glioblastoma multiforme
Time Frame: date pt started treatment to date pt last known alive
Population: latest survial data was obtained on May 30, 2006. 31/35 pts had died (89%) 21 in the +EIASD group and 10 in -EIASD group
Measure: Mean (95% Confidence Interval); unit: months
Groups:
- p450 ( +EIASD): on p450 inhibitor (Patients taking anttiseizure drugs that are known to induce the hepatic drug-metabolizing enzymes - including phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine)
  latest survial data was obtained on May 30, 2006. 31/35 pts had died (89%) 21 in the +EIASD group and 10 in -EIASD group
- nonp450 (-EIASD): not on p450 inhibitor (Patients either NOT taking anti-seizure drugs or ones that are known to not significantly influence the hepatic drug-metabolizing enzymes - including gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine,topiramate, zonisamide and filbamate.
  latest survial data was obtained on May 30, 2006. 31/35 pts had died (89%) 21 in the +EIASD group and 10 in -EIASD group
Arm/Group | p450 ( +EIASD) | nonp450 (-EIASD)
Number analyzed (Participants) | 21 | 10
months | 11.5 [8 to 16] | 16 [6 to 18]
Statistical Analysis 1: Comparison: p450 ( +EIASD) vs nonp450 (-EIASD); Test type: Non-Inferiority or Equivalence — equivalence analysis; p = 0.11, Log Rank; Hazard Ratio (HR) = 2.7, 95% CI 2-sided [1.1 to 6.3], Standard Deviation 1.8

ADVERSE EVENTS:
Time Frame: until pts progressed off treatment - in this study approximately avg 117 days.
Groups:
- P450 ARM: on p450 inhibitor (Patients taking anttiseizure drugs that are known to induce the hepatic drug-metabolizing enzymes - including phenytoin, carbamazepine, phenobarbital, primidone and oxcarbazepine)
- Non P450 ARM: NOT on p450 inhibitor *non P450 ARM (Patients either NOT taking anti-seizure drugs or ones that are known to not significantly influence the hepatic drug-metabolizing enzymes - including gabapentin, lamotrigine, valproic acid, levetiracetam, tiagabine,topiramate, zonisamide and filbamate, Keppra.
Arm/Group | P450 ARM | Non P450 ARM
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/13
Other Adverse Events (participants affected / at risk) | 22/22 | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P450 ARM (N=22) | Non P450 ARM (N=13)
abdominal pain or cramping (Gastrointestinal disorders) | 1 (2) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
ataxia (Nervous system disorders) | 3 (3) | 1 (1)
Auditory/Hearing (Ear and labyrinth disorders) | 1 (2) | 0 (0) — hearing loss
confusion (Psychiatric disorders) | 5 (5) | 1 (1)
constipation (Gastrointestinal disorders) | 4 (5) | 1 (1)
cushingoid appearance (Endocrine disorders) | 5 (6) | 5 (7)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Dizziness/lightheadedness (Nervous system disorders) | 5 (6) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
dyspepsia/heartburn (Gastrointestinal disorders) | 4 (5) | 5 (5)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
edema (General disorders) | 5 (6) | 1 (1)
fatigue (General disorders) | 7 (8) | 6 (7)
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
headache (Nervous system disorders) | 6 (7) | 4 (5)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
infection without neutropenia (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
memory loss (Nervous system disorders) | 0 (0) | 1 (1)
depression (Psychiatric disorders) | 1 (1) | 1 (1)
anxiety (Psychiatric disorders) | 2 (3) | 2 (2)
muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
neurology -cranial (Nervous system disorders) | 2 (2) | 1 (1)
neuropathy-motor (Nervous system disorders) | 5 (6) | 0 (0)
neuropathy - sensory (Nervous system disorders) | 1 (1) | 0 (0)
Salivary Gland Changes (Endocrine disorders) | 0 (0) | 1 (1)
radiation dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
speech impairment (Nervous system disorders) | 2 (2) | 1 (1)
taste disturbance (Nervous system disorders) | 0 (0) | 1 (1)
tearing (Eye disorders) | 1 (1) | 1 (1)
tremor (Nervous system disorders) | 2 (2) | 0 (0)
urinary frequency/urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
vision - blurred vision (Ear and labyrinth disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
weight gain (Investigations) | 1 (1) | 0 (0)
alkaline phosphatase (Investigations) | 5 (11) | 1 (1)
Hemoglobin / anemia (Blood and lymphatic system disorders) | 6 (8) | 2 (3)
Platelets (Investigations) | 3 (4) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (15) | 2 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Asoartate aminotransferase (SGOT) (Investigations) | 2 (2) | 1 (1)
alanine aminotransferase (SGPT) (Investigations) | 3 (6) | 2 (5)
bilirubin (Investigations) | 2 (2) | 1 (1)
white blood count (Investigations) | 4 (6) | 0 (0)
Photophobia (Nervous system disorders) | 2 (2) | 0 (0) — Neurology-Other
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Study ended early when results from another study became available documenting Temozolomide (TMZ) and radiation improved survival, we felt it was unethical to continue this study, our study did not include TMZ.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes